CLINICAL TRIAL: NCT05033197
Title: 1.1.1 Full Study Title: Impacts of Brain-Boosting Coordinated Aerobic Physical Activity Interventions on Cognition, Motor Skill Competence, Aerobic Fitness, Daily Physical Activity, and Psychological Well-beings
Brief Title: Physical Activity, Cognition, Motor Skills, and Well-beings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Weiyun Chen, Associate Professor, Director of Physical Activity and Health Lab, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00149529
Record Dates: First submitted 2021-08-17; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Motor Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This study used 2 arms, quasi experimental study design with one intervention group and one control group. The intervention group included fourth-grade students of two fourth-grade classes taught by the physical education teacher who received the coordinated-bilateral ball skills (CBBS) intervention training at each of the five elementary schools. The control group included fourth-grade students of other two fourth-grade classes taught by the physical education teacher who did not receive the CBBS intervention training at each of the five elementary schools.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBBS intervention group (Experimental): The CBBS intervention group received the 16-week intervention, including 16 CBBS lessons in basketball unit (two 40-minute lessons/week, 8 weeks) and 16 CBBS lessons in soccer unit (two 40-minute lessons/week, 8 weeks) during the 2018-2019 school year.
  Interventions: Behavioral: CBBS intervention

INTERVENTIONS:
Behavioral: CBBS intervention — The CBBS intervention group received the 16-week intervention, including 16 CBBS lessons in basketball unit (two 40-minute lessons/week, 8 weeks) and 16 CBBS lessons in soccer unit (two 40-minute lessons/week, 8 weeks) during the 2018-2019 school year.

SUMMARY:
The objective of this quasi-experimental study design was to examine effects of the coordinated-bilateral ball skills (CBBS) intervention on cognitive functions and aerobic fitness in elementary school students. The hypotheses of the study were: students in the intervention group will show a significant higher level of cognitive functions and aerobic fitness compared to the control students.

DETAILED DESCRIPTION:
Fourth-grade students at 5 elementary schools were recruited to participate. At each participating school, two fourth-grade classes were assigned to the CBBS intervention group and other two fourth-grade classes were assigned to the control group. The students in the intervention group received two, 30-min CBBS physical education (PE) lessons taught by the physical education teacher who were trained in implementation of the two CBBS lessons per week for 16 weeks. In contrast, the students in the control group received regular two PE lessons per week for 16 weeks taught by the other physical education teacher who were not be involved in the CBBS intervention training. All participating students who returned their parent/guardian' signed consent form were pre-tested and post-tested (immediately after the 16-week intervention) in cognitive functions and aerobic fitness. Descriptive statistics and linear mixed models were performed to analyze the data. All data analysis were conducted in Physical Activity and Health Lab of the School of Kinesiology at University of Michigan

ELIGIBILITY:
Inclusion Criteria:

* Being fourth-grade students in the class taught by either the intervention PE teacher or the comparison PE teacher.
* Consent/assent to participate in the study.
* Being able to complete all outcome measures without physical, cognitive, and mental constrains.

Exclusion Criteria:

* Having illness.
* Being injured.
* Having physical or mental impairment.

Ages: 9 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 347 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in D2 Test of Attention being assessed | Baseline and post-intervention test (immediately after the intervention)
  The d2 Test of Attention is a standardized paper and pencil letter-cancellation test that measures neuropsychology performance of the students in the areas of sustained and selective attention and concentration
Change in Progressive Aerobic Cardiovascular Endurance Run (PACER)® test being assessed | Baseline and post-intervention test (immediately after the intervention)
  A valid FITNESSGRAM PACER® test (15-meter version for school-aged children) was used to assess students' cardiorespiratory endurance during a PE lesson in the school gymnasium.

CONTACTS AND LOCATIONS:
Overall Officials: Weiyun Chen, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No